CLINICAL TRIAL: NCT03311191
Title: Quantifying Skin Oxygenation Properties in Normal vs Sun Exposed Skin
Acronym: SMARTevans
Status: Terminated | Type: Observational
Why Stopped: Ran out of funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Conor L Evans, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2017P000695
Record Dates: First submitted 2017-10-05; First posted 2017-10-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Healthy; Sun Exposure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Younger Women: Women ages 20-30 who are not pregnant will be painted with oxygen sensing bandage
  Interventions: Device: Measurement of skin oxygenation and oxygen consumption
- Younger Men: Men ages 20-30 will be painted with oxygen sensing bandage
  Interventions: Device: Measurement of skin oxygenation and oxygen consumption
- Older Women: Women ages 55-65 who are not pregnant will be painted with oxygen sensing bandage
  Interventions: Device: Measurement of skin oxygenation and oxygen consumption
- Older Men: Men ages 55-65 will be painted with oxygen sensing bandage
  Interventions: Device: Measurement of skin oxygenation and oxygen consumption

INTERVENTIONS:
Device: Measurement of skin oxygenation and oxygen consumption — Oxygenation properties will be measured using a transparent paint-on bandage formulation that consists of New-Skin liquid bandage, an oxygen-sensing metallo-porphyrin exhibiting bright red phosphorescence, and the green-fluorescing reference dye fluorescein.

SUMMARY:
This research study aims to determine if there are differences in oxygen consumption between chronically sun exposed and less sun exposed skin. This study uses a new imaging device that can detection oxygenation properties skin in a non-invasive manner.

DETAILED DESCRIPTION:
Sun and ultraviolet light exposure has both short term and long term effects on skin. While the short term effects, such as sunburn, are understood, chronic long-term sun exposure can cause changes to the skin that are not well characterized. One particular alteration may be how the skin consumes oxygen, a change that may be linked to biochemical alterations that have been observed in past studies. Measuring skin oxygen consumption has traditionally been difficult as the tools available have not been easy to incorporate into clinical studies. In this study, we overcome this barrier through the use of a new non-invasive oxygen-sensing device that can rapidly measure skin oxygenation properties such as oxygen consumption. This observational study will measure the oxygenation properties of both chronically sun exposed and less sun exposed skin in the predefined groups of both young and older men and women.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age groups: 20 - 30 and 55 - 65
* Fitzpatrick skin types I, II, III, and IV

Exclusion Criteria:

* Fitzpatrick skin types V and above
* Tattoo markings anywhere on the arm(s)
* Significant scarring or discoloration (e.g. birthmarks) on the arm(s)
* Any current injuries, infections or wounds on the arm(s)
* Routinely (4+ doses per week) take high dosages of anti-inflammatory drugs (e.g. aspirin, ibuprofen, corticosteroids), immunosuppressive drugs, or antihistamine medications. However steroid nose drops and/or eye drops are permitted.
* Has taken an anti-inflammatory drug (e.g. aspirin) within the prior 24 hours of the study visit.
* Have diabetes that is treated with injectable or oral insulin
* Have any other active or chronic skin problems on the arms
* Are currently participating in another skin care product study at this or any other facility
* Have participated in any type of skin product treatment study within the past 2 weeks
* Have or ever have had dermatographia
* Pregnant women
* Lactating women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is designed to gather data from two different age groups of men and women to evaluate the differences in skin oxygen properties, if any, between chronically sun exposed and less sun exposed skin. This study makes use of an oxygen sensing bandage device that can quantitatively measure both tissue oxygen partial pressure and oxygen consumption rate. Due to its early stage in development, the device has not yet been designed to control for high melanin content of skin. Thus only subjects with lower melanin content (i.e. Fitzpatrick skin types I - IV) will be included in the study. In addition, tattoo markings, scarring or significant natural discolorations can interfere with the imaging results by absorbing blue light and subjects with any of these will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Differences in the relative (sun exposed vs nonexposed) and absolute oxygen properties within an individual and between the two age groups | 20 min estimated per subject
  The skin's partial pressure of oxygen and oxygen consumption rate is measured at 4 different locations on the subjects arms using the oxygen sensing device, where it is expected that that difference between more sun exposed regions and less sun exposed regions will be greater in the population of older adults.

SECONDARY OUTCOMES:
The differences in the relative (sun exposed vs nonexposed) and absolute oxygen properties between the sexes | 20 min estimated per subject
  The skin's partial pressure of oxygen and oxygen consumption rate is measured using the oxygen sensing device and compared between the sexes (arm 1+3 and arm 2+4)

OTHER OUTCOMES:
The oxygen properties connected to lifestyle choices, such as sun-seeking behavior, lifetime sun exposure levels, and smoking. | 20 min estimated per subject, plus time to fill in questionnaire response
  The skin's partial pressure of oxygen and oxygen consumption rate is measured with the oxygen sensing device and compared between groups stratified by lifestyle, as based on subject responses from the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Conor L Evans, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
This study was funded by a research gift from Procter & Gamble. While the investigator is under no obligation to do so, research results and/or study data may be shared with the company for purposes of future scientific publications and/or research collaborations. However, information shared with the company will not include any identifiers that could be used to link data to individual subjects.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As collected; until the study is complete and the results and published.
Access Criteria: Image data files and subject questionnaires may be used after the study for future research. However, no individually identifiable patient information will be correlated with or otherwise used with the study data. Specimens and data will not be stored at collaborating sites outside of Partners Healthcare.

REFERENCES:
- [Background] Koolen PGL, Li Z, Roussakis E, Paul MA, Ibrahim AMS, Matyal R, Huang T, Evans CL, Lin SJ. Oxygen-Sensing Paint-On Bandage: Calibration of a Novel Approach in Tissue Perfusion Assessment. Plast Reconstr Surg. 2017 Jul;140(1):89-96. doi: 10.1097/PRS.0000000000003421. PMID 28654595
- [Background] Roussakis E, Li Z, Nowell NH, Nichols AJ, Evans CL. Bright, "Clickable" Porphyrins for the Visualization of Oxygenation under Ambient Light. Angew Chem Int Ed Engl. 2015 Dec 1;54(49):14728-31. doi: 10.1002/anie.201506847. Epub 2015 Oct 29. PMID 26510549
- See also: Recruitment Link — https://clinicaltrials.partners.org/study/smartevans